CLINICAL TRIAL: NCT05556226
Title: A Phase 1 Study in Healthy Subjects to Evaluate the Relative Bioavailability of ABBV-154
Brief Title: Study to Assess Adverse Events and Compare How Two Subcutaneous ABBV-154 Injection Formulations Move Through the Body of Adult Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M23-506
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: ABBV-154
Keywords: ABBV-154

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABBV-154 Dose A (Experimental): Participants will receive subcutaneous dose of ABBV-154 Dose Formulation A.
  Interventions: Drug: ABBV-154 Dose Formulation A
- ABBV-154 Dose B (Experimental): Participants will receive subcutaneous dose of ABBV-154 Dose Formulation B.
  Interventions: Drug: ABBV-154 Dose Formulation B

INTERVENTIONS:
Drug: ABBV-154 Dose Formulation A — Subcutaneous Injection
  Arms: ABBV-154 Dose A
Drug: ABBV-154 Dose Formulation B — Subcutaneous Injection
  Arms: ABBV-154 Dose B

SUMMARY:
This study will assess how safe ABBV-154 is and how ABBV-154 moves through the body of adult healthy participants. Adverse Events will be assessed.

ABBV-154 is an investigational drug being developed for potential treatment of immune-mediated inflammatory diseases. Participants are randomly assigned to one of the 2 treatment groups. Approximately 40 adult healthy volunteers will be enrolled in 2 sites in the United States.

All participants will receive ABBV-154 as subcutaneous injections with one of the 2 different formulations.

There may be higher burden for participants in this trial. Participants will be confined for 9 days. Adverse Events and blood tests will be performed.

ELIGIBILITY:
Inclusion Criteria:

- Body Mass Index (BMI) is ≥ 18.0 to ≤ 29.9 kg/m2 after rounding to the nearest tenth at screening and upon initial confinement.

Exclusion Criteria:

* Participant using any medications, vitamins and/or herbal supplements, within the 2 week period or 5 half-lives (whichever is longer) prior to study drug administration.
* History of epilepsy, any clinically significant cardiac, respiratory (except mild asthma), renal, hepatic, gastrointestinal, hematologic, demyelinating disease (including myelitis) or neurologic symptoms suggestive of demyelinating disease, glaucoma, psychiatric disease or disorder, or any uncontrolled medical illness.
* Prior exposure to similar biologic therapies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Approximately up to 58 days
  Maximum Observed Plasma Concentration (Cmax)
Time to Maximum Observed Plasma Concentration (Tmax) | Approximately up to 58 days
  Time to Maximum Observed Plasma Concentration (Tmax)
Apparent Terminal Phase Elimination Rate Constant (β) | Approximately up to 58 days
  Apparent Terminal Phase Elimination Rate Constant (β)
The Terminal Phase Elimination Half-Life (t1/2) | Approximately up to 58 days
  The Terminal Phase Elimination Half-Life (t1/2)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt) | Approximately up to 58 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Time of the Last Measurable Concentration (AUCt)
The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞) | Approximately up to 58 days
  The Area Under the Plasma Concentration-Time Curve (AUC) from Time 0 to Infinity (AUC∞)
Number of Participants with Adverse Events | Approximately up to 72 days
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Acpru /Id# 250429, Grayslake, Illinois
  - PPD Clinical Research Unit -Las Vegas /ID# 250650, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: No